CLINICAL TRIAL: NCT03543605
Title: Impacto clínico y microbiológico de un Programa de optimización de Antimicrobianos específico Para Centros Socio-sanitarios. Ensayo clínico Aleatorizado Por Grupos. Ensayo PROA-SENIOR
Brief Title: Clinical/Microbiological Impact of a Specific Antimicrobial Stewardship Program for Nursing Homes
Acronym: PROA-SENIOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PROA-SENIOR (PRO-FIS-2017-01)
Record Dates: First submitted 2018-05-08; First posted 2018-06-01 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Human Microbiome; Antibiotic Resistant Infection; Nursing Homes

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The study will be masked in the first year (pre-intervention) and open in the year of intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PROA Experimental (Experimental): It consists of the intervention measures described in the general antimicrobial stewardship program (PROA Control) plus clinical advice.
  * The clinical assessments have been adapted for this project to the unique characteristics of infectious diseases in nursing homes.
  * These are individual training activities whose main objective is to modify prescribing behaviors when they are inadequate and reinforce them when they are correct.
  * They are carried out between the medical adviser, an expert in infectious diseases, and the doctor of the nursing home, through the structured review of a case attended by the doctor in the last 24 hours. The recommendations are not compulsory, and do not seek to change the decisions made in that patient, but the future ones in the case that is necessary.
  * The counseling will be done by video-conference, with an approximate duration of 10 minutes. Each of the doctors will receive two monthly assessments during the intervention period.
  Interventions: Behavioral: PROA Experimental
- PROA Control (Other): The intervention of the general antimicrobial stewardship program (PROA) contains the following set of measures:
  * Creation of the local team of the PROA: one of the Family Physicians responsible for the patients and the pharmacist of the reference hospital of the center.
  * Presentation of the project by the local team in its own center.
  * Choice of the Aljarafe guide as a reference document for the diagnosis and treatment of infectious diseases. It is an accredited guide and widely disseminated among primary care and hospital doctors.
  * Permanent information of the project (poster with its synthesis, a pocket triptych with the guide for the clinical management of the main clinical syndromes of infections in the residents of the nursing homes).
  * Feedback of the results that will serve each center to know the evolution of its results, and to stimulate the comparison with the other centers.
  Interventions: Other: PROA Control

INTERVENTIONS:
Behavioral: PROA Experimental — PROA Control plus clinical advice
  Arms: PROA Experimental
Other: PROA Control — PROA Control
  Arms: PROA Control

SUMMARY:
Background: In nursing homes, excessive and inappropriate use of antimicrobials, adverse events caused by these drugs, and infections by multidrug-resistant bacteria (MDRB) are more frequent than in the general population, posing a serious Public Health risk. Antimicrobial stewardship programs (ASP) are a key strategy to improve the use of antibiotics and to fight against bacterial resistance. Its usefulness in hospitals has been demonstrated. The Centers for Disease Control and Prevention urge the implementation ASP in nursing homes, with measures taken from the ASP in hospitals, but the available information is so limited that it does not allow specific recommendations to be made for these centers.

Objectives: To know if an ASP with an individual intervention measure, the clinical assessments, is better to an ASP with general intervention measures, both designed specifically for nursing homes, and what is the clinical and ecological impact of both, on the baseline situation.

Methods: a) Randomized clinical trial, in parallel groups, for comparison of both ASP. b) Quasi-Experimental study of timeseries for the evaluation of the clinical and ecological impact on the baseline situation. The following indicators will be analyzed: the use of antimicrobials in the centers; the intestinal microbiota diversity of nursing home residents, and the incidence of MDRB and Clostridium difficile infections; and the frequency of adverse events caused by antimicrobials and hospital admissions for infections. The study population will be 2.220 residents from 20 public nursing homes.

ELIGIBILITY:
Inclusion Criteria:

* Public nursing homes under the ownership of the Department of Equality and Social Policies of the Junta de Andalucía

Exclusion Criteria:

* Nursing homes that are not under the ownership of the Department of Equality and Social Policies of the Junta de Andalucía

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1667 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change of Total antimicrobial pressure | From date of randomization, assessed monthly up to 12 months
  Change from baseline of antimicrobial pressure, which will be measured using the recommended international standard, the defined daily dose (DDD) / 1000 residents / day

SECONDARY OUTCOMES:
Antimicrobials adverse events | From date of randomization, assessed monthly up to 12 months
  The frequency of side effects of the antimicrobials that require admission will be evaluated by measuring the number of hospital admissions due to adverse effects of antimicrobials / 1000 residents / day.
Incidence of infections by multiresistant bacteria | From date of randomization, assessed monthly up to 12 months
  Incidence density (number of isolates in clinical samples / 1000 residents / day) of the following pathogens: quinolone resistant E.coli; E. coli BLEE, Klebsiella pneumoniae BLEE, carbapenemase-producing enterobacteria, methicillin-resistant Staphylococcus aureus (MRSA), in samples sent for culture.
Incidence of infections of C. difficile | From date of randomization, assessed monthly up to 12 months
  Incidence density (number of C. difficile isolates in clinical samples / 1000 residents / day) sent for toxin detection.

CONTACTS AND LOCATIONS:
Overall Officials: José Miguel Cisneros Herreros, PhD, MD, Principal Investigator — Virgen del Rocío University Hospital
Locations (1):
- Virgen del Rocío University Hospital, Seville, Spain

REFERENCES:
- [Derived] Penalva G, Crespo-Rivas JC, Guisado-Gil AB, Rodriguez-Villodres A, Pachon-Ibanez ME, Cachero-Alba B, Rivas-Romero B, Gil-Moreno J, Galva-Borras MI, Garcia-Moreno M, Salamanca-Bautista MD, Martinez-Rascon MB, Cantudo-Cuenca MR, Ninahuaman-Poma RC, Enrique-Miron MLA, Perez-Barroso A, Marin-Ariza I, Gonzalez-Florido M, Mora-Santiago MDR, Belda-Rustarazo S, Exposito-Tirado JA, Rosso-Fernandez CM, Gil-Navarro MV, Lepe-Jimenez JA, Cisneros JM; PROA-SENIOR Study Group. Clinical and Ecological Impact of an Educational Program to Optimize Antibiotic Treatments in Nursing Homes (PROA-SENIOR): A Cluster, Randomized, Controlled Trial and Interrupted Time-Series Analysis. Clin Infect Dis. 2023 Mar 4;76(5):824-832. doi: 10.1093/cid/ciac834. PMID 36268822